CLINICAL TRIAL: NCT01041768
Title: Multicentric Prospective Randomized Controlled Trial on the Effect of Gastric Bypass and Bilopancreatic Diversion on Type 2 Diabetes Mellitus in Patients With BMI Between 30 and 35
Brief Title: Multicentric Prospective Randomized Trial on Surgery Versus Standard Medical Care in Type 2 Diabetic Patients BMI 30-35
Acronym: DIA-CHIR-MULT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: IRCCS Azienda Ospedaliera Universitaria San Martino - IST Istituto Nazionale per la Ricerca sul Cancro, Genoa, Italy (Other)
Collaborators: Ospedale di Desenzano del Garda (Unknown); Azienda Ospedaliero, Universitaria Pisana (Other); Azienda Ospedaliera Santa Maria Degli Angeli (Other); IRCCS Multimedica (Other); Istituto Clinico Humanitas (Other); Ospedale Polispecialistico Humanitas Gavazzeni, Bergamo (Unknown); Azienda Sanitaria Locale n. 2 - Lanciano Vasto Chieti (Other); Ente Ospedaliero Ospedali Galliera (Other); Ospedale S. Giovanni Bosco (Other); Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other); University of Rome Tor Vergata (Other); Azienda Ospedaliera San Giovanni Battista (Other); Ospedale S. Timoteo, Termoli (Unknown); Ospedale Marino, Cagliari (Unknown); Hospital San Pietro Fatebenefratelli (Other); Azienda Ospedaliera Universitaria Policlinico (Other); Azienda ospedaliera Garibaldi Catania (Unknown)
Responsible Party: Nicola Scopinaro, Prof., Azienda Ospedaliera Universitaria "San Martino"
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DIA-CHIR-MULT-BMI 30-35
Record Dates: First submitted 2009-12-31; First posted 2010-01-01 (Estimated); Last update posted 2010-03-30 (Estimated); Status verified 2009-12

CONDITIONS: Diabetes Mellitus
Keywords: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — Bariatric Surgery; Biliopancreatic Diversion; Gastric Bypass

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- antidiabetic medical therapy (Active Comparator)
  Interventions: Procedure: Bariatric surgery
- Bariatric Surgery (Experimental)
  Interventions: Procedure: Bariatric surgery

INTERVENTIONS:
Procedure: Bariatric surgery — Biliopancreatic diversion consists of a distal gastrectomy with a long Roux-en-Y reconstruction, where the enteroenterostomy is placed 50 cm proximal to the ileocecal valve; Gastric bypass consists of creating a small proximal gastric pouch by division of the upper stomach, with reconstruction of the GI continuity by means of a Roux-en-Y loop
  Other Names: biliopancreatic diversion; gastric bypass

SUMMARY:
200 type 2 diabetic patients -BMI between 30-35- will be submitted to bariatric surgery (biliopancreatic diversion BPD or gastric bypass GBP ) and 100 will receive standard medical treatment.

Subjects will be monitored during a 5 year period to assess the effects of the surgical procedures on diabetes resolution and control at 1, 3 and 5 years.

DETAILED DESCRIPTION:
The study is a multicentric prospective 2-arm randomized controlled trial. Only Centers with at least 50 bariatric surgeries performed during the time window January 2007 and September 2008 will be allowed to participate in the study.

Each Collaborating Center participating in the study will perform only one type of surgical procedure (GBP or BPD), depending on which one it is more familiar with.

Patients will be randomly assigned with a 2 to 1 ratio to receive either bariatric surgery (BS) (either GBP or BPD) or standard antidiabetic care (AC). The randomization will be centralized in the Coordinating Center. Patients assigned to BS will undergo GBP or BPD, depending on each Collaborating Center. Recruitment will continue, independently of the number of recruited patients per center, until the target of 200 GBP+BPD patients, and 100 AC patients will be attained.

After one year since enrollment, patients in AC group will be offered the choice to undergo one of the two surgical procedures, and then will follow the same protocol study as the other surgical patients. In addition, each Collaborating Center will be responsible for selecting one diabetic subject for each operated patient, matched as closely as possible with the patients assigned to surgical therapy, from the local population in medical treatment. These patients will serve as controls for long term mortality and morbidity.

ELIGIBILITY:
Inclusion Criteria:

* BMI ≥30 and ≤34.9 kg/m2
* age between 35 and 70 years
* duration of diabetes ≥ 5 years
* poor glycemic control (i.e., HbA1c ≥ 8%) in spite a medical antidiabetic therapy in accordance with good clinical practice (GCP)
* presence of significant co-morbidities or complications (such as dyslipidemia, arterial hypertension, impaired renal function, neuropathy, retinopathy, CVD)

Exclusion Criteria:

* specific contraindication to obesity surgery or GBP or BPD, including any gastric alteration specifically contraindicating GBP
* HbA1c < 8%
* positive autoantibodies anti-pancreas islet
* serum C-peptide < 0.5 ng/ml
* pregnancy
* medical conditions requiring acute hospitalisation
* severe diabetes complications or associated medical conditions (such as blindness, end-stage renal failure, liver cirrhosis, malignancy, chronic congestive heart failure
* recent (within preceding 12 months) myocardial infarction, stroke or TIA
* unstable angina pectoris
* psychological conditions which may hamper patient's cooperation
* geographic inaccessibility
* any condition which, in the judgement of the Investigator, may make risky the participation in the study or bias the results

Ages: 35 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2009-03; Primary Completion 2010-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients achieving diabetes complete remission (HbA1c 6% or below) or diabetes control (HbA1c between 7% and 6.1%) on free diet and with no antidiabetic medical therapy. | year 1, 3, 5

SECONDARY OUTCOMES:
Stable reduction of preoperative HbA1c; BMI; mortality/morbidity; Major components of the metabolic syndrome; Diabetes complications; Improvement of beta-cell function; insulin resistance reduction ; Overall and CV disease mortality. | at and post surgery, 1,3, 5 years since randomization

CONTACTS AND LOCATIONS:
Overall Officials: Nicola Scopinaro, MD, Principal Investigator — Azienda Ospedaliera Universitaria "San Martino", Genova, Italy
Locations (1):
- Azienda Ospedaliera Universitaria "San Martino", Genova, Italy